CLINICAL TRIAL: NCT00810797
Title: Intermittent Exemestane Therapy for Metastatic Breast Cancer
Brief Title: Exemestane in Treating Postmenopausal Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08063; P30CA033572 (NIH); CHNMC-08063; CDR0000629864 (Registry Identifier: NCI PDQ); NCI-2010-00761 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (exemestane) (Experimental): Patients receive oral exemestane once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: exemestane; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: exemestane — Given orally
Other: laboratory biomarker analysis — One year after completion of study treatment
Procedure: quality-of-life assessment — One year after completion of study treatment
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by lowering the amount of estrogen the body makes.

PURPOSE: This phase II trial is studying how well exemestane works in treating postmenopausal women with stage IV breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression-free survival at 4 months, as measured by Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OBJECTIVES:

I. Objective response rate (complete response [CR] and partial response [PR]).

II. Clinical benefit (CR, PR, and stable disease >= 6 months).

III. Assessment of toxicity.

IV. Assessment of compliance with medication adherence.

V. Assessment of quality of life.

VI. Assessment of bone health.

TERTIARY OBJECTIVES:

I. Serial measurements of serum estradiol, estrone, and estrone sulfate.

II. To investigate treatment resistance (e.g., expression of amphiregulin, epidermal growth factor receptor [EGFR]), using molecular and immunohistochemical analyses of blood and tumor samples of pre- and post- (when available) treatment tissues. Microarray analyses to quantitate the expression of specific estrogen-responsive genes (e.g. thyroid transcription factor 1 [TTF1] and PDZK1) will also be performed.

OUTLINE: Patients receive exemestane orally (PO) once daily (QD) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic carcinoma of the breast
* Hormone receptor (estrogen receptor [ER] and/or progesterone receptor [PR]) positive disease (defined as: ER and/or PR positivity as >= 5% staining), as confirmed by immunohistochemistry (IHC) based on primary breast tissue or metastatic tissue
* Postmenopausal, as defined by any of the following:
* Natural menopause, with at least 1 year since last menses
* Chemotherapy-induced menopause with at least 1 year from last menses and serum luteinizing hormone (LH)/follicle-stimulating hormone (FSH) and estradiol levels within the postmenopausal range
* History of surgical or radiation-induced ovarian ablation
* For women =< 56 years old and with a history of hysterectomy but at least one ovary intact, serum LH/FSH and estradiol levels must be within the postmenopausal range
* Postmenopausal women with disease recurrence while receiving either tamoxifen or a non-steroidal aromatase inhibitor (AI) as adjuvant therapy (as long as adjuvant hormonal therapy was taken for 6 months before disease progression) or with disease recurrence following the discontinuation/completion of adjuvant hormonal therapy
* Postmenopausal women with disease progression following either 0, 1 or 2 prior hormonal therapies for metastatic breast cancer, as long as the subject has had no prior exposure to exemestane (EXE)
* Measurable or non-measurable (but evaluable) disease, as defined by RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Neutrophil count >= 1.5 X 10^9 cells/L
* Platelet count >= 100 X 10^9 cells/L
* Serum creatinine =< 1.5 times upper limit of normal (ULN)
* Total serum bilirubin =< 1.5 times ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) levels =< 2.5 x ULN in patients without liver metastases or =< 5 times ULN in patients with liver metastases
* Alkaline phosphatase =< 2.5 times the ULN for patients without bone or liver metastases
* Subjects must have an estimated life expectancy of greater than 6 months

Exclusion Criteria:

* Prior exposure to EXE, whether in the adjuvant or metastatic setting
* Prior history of any other cancer with the exception of non-melanoma skin cancer and treated in situ carcinoma of the cervix
* Active or symptomatic central nervous system (CNS) metastasis (stable or treated brain metastasis allowed but patients must be off decadron, if given for CNS disease)
* Hormone-receptor negative or unknown breast cancer
* More than two prior chemotherapy regimen for treatment of metastatic disease (any prior chemotherapy given in the adjuvant setting is permitted)
* Administration of any other anti-cancer therapy within 2 weeks of initiating study treatment; use of bisphosphonates, however, are permitted for patients with known bone metastases
* Treatment with any other concurrent investigational agent or anti-tumor drug (chemotherapy, antibody therapy or other biologic agents), will not be permitted
* Subjects who have had no prior exposure to endocrine therapy
* Any uncontrolled medical co-morbidity or psychiatric disorder which interferes with the ability to provide informed consent or comply with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12-02; Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Exemestane): Patients receive 25mg oral exemestane once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  exemestane: Given orally
  laboratory biomarker analysis: One year after completion of study treatment
  quality-of-life assessment: One year after completion of study treatment
  immunohistochemistry staining method: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Exemestane)
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 60 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13
  Hispanic | 15
  African American | 1
  Asian | 4
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Until disease progression of death from any cause, up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 36
months | 4.3 [2.0 to 6.5]

2. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Until disease progression or off treatment, assessed up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 36
percentage of participants | 8.3 [1.8 to 22.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 5 years and 8 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Exemestane)
All-Cause Mortality (participants affected / at risk) | 30/36
Serious Adverse Events (participants affected / at risk) | 4/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Exemestane) (N=36)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Exemestane) (N=36)
Hemoglobin decreased (Blood and lymphatic system disorders) | 18 (89)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (4)
Palpitations (Cardiac disorders) | 2 (4)
Pericardial effusion (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (15)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (4)
Vision blurred (Eye disorders) | 2 (5)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (21)
Constipation (Gastrointestinal disorders) | 13 (28)
Diarrhea (Gastrointestinal disorders) | 11 (39)
Dry mouth (Gastrointestinal disorders) | 2 (7)
Dyspepsia (Gastrointestinal disorders) | 6 (8)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 7 (8)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (55)
Oral pain (Gastrointestinal disorders) | 5 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 2 (4)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)
Chest pain (General disorders) | 5 (5)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 9 (37)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 20 (107)
Fever (General disorders) | 6 (10)
Gait abnormal (General disorders) | 1 (1)
Ill-defined disorder (General disorders) | 2 (4)
Irritability (General disorders) | 5 (20)
Localized edema (General disorders) | 2 (3)
Pain (General disorders) | 14 (52)
Bronchitis (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative gastrointestinal injury - Oral cavity NOS (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 9 (17)
Alkaline phosphatase increased (Investigations) | 13 (70)
Aspartate aminotransferase increased (Investigations) | 21 (56)
Bilirubin increased (Investigations) | 4 (18)
Coagulopathy (Investigations) | 1 (1)
Creatine phosphokinase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 5 (41)
Haptoglobin decreased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 11 (29)
Lymphocyte count decreased (Investigations) | 6 (16)
Neutrophil count decreased (Investigations) | 7 (18)
Platelet count decreased (Investigations) | 9 (19)
Serum cholesterol increased (Investigations) | 1 (1)
Weight gain (Investigations) | 4 (15)
Weight loss (Investigations) | 3 (13)
Anorexia (Metabolism and nutrition disorders) | 8 (29)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 22 (120)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (8)
Serum calcium increased (Metabolism and nutrition disorders) | 10 (24)
Serum glucose decreased (Metabolism and nutrition disorders) | 7 (10)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 8 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 13 (26)
Serum sodium increased (Metabolism and nutrition disorders) | 5 (7)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (36)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (51)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Fibrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 16 (111)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (28)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 5 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (34)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (43)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Cognitive disturbance (Nervous system disorders) | 2 (6)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (8)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (36)
Memory impairment (Nervous system disorders) | 5 (44)
Peripheral motor neuropathy (Nervous system disorders) | 4 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (26)
Tremor (Nervous system disorders) | 2 (3)
Trigeminal nerve disorder (Nervous system disorders) | 1 (2)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 11 (36)
Confusion (Psychiatric disorders) | 3 (8)
Depression (Psychiatric disorders) | 9 (27)
Insomnia (Psychiatric disorders) | 11 (46)
Libido decreased (Psychiatric disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (2)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 2 (3)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (21)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (30)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (19)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Sweating (Skin and subcutaneous tissue disorders) | 5 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 24 (105)
Hypertension (Vascular disorders) | 5 (16)
Hypotension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT00810797/Prot_SAP_000.pdf